CLINICAL TRIAL: NCT06358001
Title: EchoTip AcuCore Post-Market Clinical Study
Status: Completed | Type: Observational
Sponsor: Cook Research Incorporated (Industry)
Responsible Party: Sponsor
Organization: Cook Group Incorporated (Industry)
Other Study IDs: 21-07
Record Dates: First submitted 2024-04-05; First posted 2024-04-10 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Adenocarcinoma; Neuroendocrine Tumors; Hepatocellular Carcinoma; Cholangiocarcinoma; Malignant Lymphoma; Metastasis; Chronic Pancreatitis; Autoimmune Pancreatitis
Keywords: Fine needle biopsy (FNB); Core biopsy; Endoscopic ultrasonography-guided fine-needle biopsy (EUS-FNB); Tissue Diagnosis; Histology; Endoscopic ultrasound; Interventional EUS; Pancreas
MeSH Terms: conditions — Adenocarcinoma; Neuroendocrine Tumors; Carcinoma, Hepatocellular; Cholangiocarcinoma; Lymphoma; Neoplasm Metastasis; Pancreatitis, Chronic; Autoimmune Pancreatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- EchoTip AcuCore: Patients with use of AcuCore 22 gauge FNB to collect specimens from GI tract
  Interventions: Device: EchoTip AcuCore

INTERVENTIONS:
Device: EchoTip AcuCore — Using endoscopic ultrasound guided needle to collect biopsies

SUMMARY:
The purpose of collecting this data is to continue to learn more about the EchoTip AcuCore and the device's ability to produce the desired favorable effect and if there are any undesired outcomes that may be related to the EchoTip AcuCore.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been referred for an endoscopic ultrasound (EUS) fine needle biopsy procedure
* The EchoTip AcuCore device is the first EUS biopsy needle used in the procedure.

Exclusion Criteria:

* Patient's age is less than 18 years
* Patient is unable or unwilling to sign and date the informed consent. If IRB approves a waiver of consent, this exclusion criterion is not applicable.
* Patient is simultaneously participating in another pre-market investigational drug or pre-market investigational device study involving an EUS fine needle biopsy procedure and for which the patient has not completed the follow-up phase for the primary endpoint at least 30 days prior to enrollment in this study.
* Inaccessible or unsuitable lesion (lesion not visualized or a large vessel, duct or primary mass interposition)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients referred for a EUS-FNB procedure will be considered for enrollment
Sampling Method: Non-Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2024-08-05 (Actual); Primary Completion 2025-06-14 (Actual); Study Completion 2025-07-19 (Actual)

PRIMARY OUTCOMES:
Technical Success | Duration of the procedure (approx. 1 hr)
  The ability to obtain a sample without failure of the needle system necessitating the use of a new needle to complete the procedure

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - University of California, Irvine, Orange, California
  - Advent Health, Porter, Denver, Colorado
  - Shands Hospital-University of Florida, Gainesville, Florida
  - University of Florida Shands Hospital, Gainesville, Florida
  - Advent Health Medical Group, Orlando, Orlando, Florida
  - Geisinger Medical Center, Danville, Pennsylvania
  - University of Texas Memorial Hermann Hospital, Houston, Texas
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Undecided
Cook Research Incorporated (CRI) is fully committed to supporting the principles of responsible data sharing, including providing qualified scientific researchers access to deidentified, patient-level data from CRI clinical studies to conduct legitimate scientific research. Data underlying the results reported in this clinical study will be made available for request immediately after approval or clearance of the product and ending 5 years after approval or clearance. Interested researchers may review the "Cook Research Incorporated Policy on Access to Clinical Study Data" at https://www.cookresearchinc.com/extranet/data-access.html and submit a complete research proposal to request data access. Additional study documents (such as the study protocol) will be shared as needed if the data access request is granted. A data sharing agreement will be executed for access to deidentified patient-level data.